CLINICAL TRIAL: NCT02918981
Title: Nutritional Strategies to Augment the Postprandial Muscle Protein Synthetic Response to the Ingestion of a Low Dose of Protein in Middle-aged Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Urbana-Champaign (Other)
Responsible Party: Principal Investigator, Nicholas Burd, Assistant Professor, University of Illinois at Urbana-Champaign
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 16999
Record Dates: First submitted 2016-09-20; First posted 2016-09-29 (Estimated); Last update posted 2020-11-03 (Actual); Status verified 2020-11

CONDITIONS: Aging
MeSH Terms: interventions — Resistance Training; Whey Proteins; Leucine; Citrulline

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Whey protein (Active Comparator): After resistance exercise, participants aged 50-79 years will consume 14g Whey protein dissolved in 200 mL of water
  Interventions: Behavioral: Resistance Exercise; Dietary Supplement: 14 g Whey protein
- Whey + Leucine (Experimental): After resistance exercise, participants aged 50-79 years will consume 6.6 g Whey protein + 1.25 g Leucine dissolved in 200 mL of water
  Interventions: Behavioral: Resistance Exercise; Dietary Supplement: 6.6 g Whey protein + 1.25 g leucine
- Whey + Leucine + Whey peptides (Experimental): After resistance exercise, participants aged 50-79 years will consume 4 g Whey protein + 1.25 g Leucine + 2.6 g Whey peptides dissolved in 200 mL of water
  Interventions: Behavioral: Resistance Exercise; Dietary Supplement: 4 g Whey protein + 1.25 g leucine + 2.6 g Whey peptides
- Whey + Leucine + Citrulline (Experimental): After resistance exercise, participants aged 50-79 years will consume 6.6 g Whey protein + 1.25 g Leucine + 0.8 g Citrulline dissolved in 200 mL of water
  Interventions: Behavioral: Resistance Exercise; Dietary Supplement: 6.6 g Whey protein + 1.25 g leucine + 0.8 g Citrulline
- Water (Sham Comparator): After resistance exercise, participants aged either 20-30 or 50-79 years old will consume 200 mL water
  Interventions: Behavioral: Resistance Exercise; Other: Water control

INTERVENTIONS:
Behavioral: Resistance Exercise — Participants will perform unilateral leg extension exercise immediately prior to ingestion of the experimental beverage
Dietary Supplement: 14 g Whey protein
  Arms: Whey protein
Dietary Supplement: 6.6 g Whey protein + 1.25 g leucine
  Arms: Whey + Leucine
Dietary Supplement: 4 g Whey protein + 1.25 g leucine + 2.6 g Whey peptides
  Arms: Whey + Leucine + Whey peptides
Dietary Supplement: 6.6 g Whey protein + 1.25 g leucine + 0.8 g Citrulline
  Arms: Whey + Leucine + Citrulline
Other: Water control
  Arms: Water

SUMMARY:
Using stable isotope methodology, investigators will determine the postabsorptive and postprandial muscle protein synthetic response in 60 female adults (Age 50-79, BMI: <30 kg/m2) immediately after an acute bout of resistance exercise. Participants will be divided in to 5 groups of twelve women (n=12). Each group will receive a different protein beverage or placebo to consume following the resistance exercise training. Group 1 will consume a beverage consisting of whey protein; group 2 will consume whey protein supplemented with additional leucine; group 3 will consume whey protein supplemented with additional leucine and hydrolyzed whey peptides; group 4 will consume whey protein supplemented with additional leucine and citrulline; group 5 will just consume water. During the testing, blood and muscle samples will be collected.

ELIGIBILITY:
Inclusion Criteria:

* BMI <30 kg/m2
* Healthy, sedentary
* Either 20-30 years old or 50-79 years old

Exclusion Criteria:

* Tobacco use
* Allergies to milk consumption
* Unusually high protein consumption
* Vegan diet
* Allergies to antibiotics or xylocaine
* Phenylketonuria (PKU)
* Diagnosed GI tract diseases
* Arthritic conditions
* A history of neuromuscular problems
* Heart disease
* Metabolic disorders
* -Liver, kidney, or urinary disease
* Musculoskeletal problems
* Autoimmune disease
* Neurological disease
* Previous participation in amino acid tracer studies
* Predisposition to hypertrophic scarring or keloid formation
* Individuals on any medications known to affect protein metabolism (i.e. corticosteroids, non-steroidal anti-inflammatories, or prescription strength acne medications).
* Individuals using thyroid medications or other medications affecting endocrine function
* Pregnancy
* Contraindications for exercise
* BMI ≥30
* supplements that influence protein metabolism (e.g omega 3 fish oils)

Ages: 20 Years to 79 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2019-03-06 (Actual); Study Completion 2019-03-06 (Actual)

PRIMARY OUTCOMES:
The myofibrillar protein synthetic response to protein ingestion | Postabsorptive for 3 hours, Postprandial for 4 hours hours
  Myofibrillar protein synthesis rates will be assessed during the postabsorptive period for 3 hr and during the 4 hr after the ingestion of the experimental beverages. This will allow us to assess the change from the postabsorptive to the postprandial period

SECONDARY OUTCOMES:
mTORC1 phosphorylation | Baseline and at 2 and 4 hours after protein ingestion
  Activation of anabolic signaling pathways will be assessed in the fasted state and at 2 and 4 hr after the ingestion of the experimental beverages.

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas A Burd, Ph.D., Principal Investigator — University of Illinois at Chicago
Locations (1):
- Freer Hall, Urbana, Illinois, United States

IPD SHARING:
Plan to Share IPD: No